CLINICAL TRIAL: NCT00228813
Title: Feasibility Study of Using G-CSF Stimulated Bone Marrow and In Vivo T-Cell Depletion in Patients With Hematologic Malignancies or Bone Marrow Failure Syndrome With Partially Mismatched Related Donors
Brief Title: G-CSF PMRD: Granulocyte Colony Stimulating Factor (G-CSF) Stimulated Bone Marrow and In Vivo T-Cell Depletion in Patients With Hematologic Malignancies or Bone Marrow Failure Syndrome
Acronym: G-CSF PMRD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of enrollment
Sponsor: Emory University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00021819; 0159-2004 (Other: Emory University)
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Results first posted 2016-07-06 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-08

CONDITIONS: Hematologic Malignancies
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Granulocyte Colony Stimulating Factor (G-CSF) stimulation (Other): Participants will receive bone marrow from donors who undergo Granulocyte Colony Stimulating Factor (G-CSF) stimulation prior to bone marrow collection.
  Interventions: Drug: Granulocyte Colony Stimulating Factor

INTERVENTIONS:
Drug: Granulocyte Colony Stimulating Factor — FILGRASTIM: G-CSF (NEUPOGEN®) is administered as a short IV infusion over 30 minutes or subcutaneously. It is given beginning on day -3 for 3 days to the donor prior to the bone marrow harvest.
  Drug Information: FILGRASTIM: G-CSF (Neupogen®) Formulation: G-CSF is available as a preservative-free solution for injection in 1.0 ml and 1.6 ml vials containing 300 mcg/ml.
  Administration: G-CSF 5 mcg/kg/d will be given subcutaneously or as a short I.V. infusion over 30 minutes.
  Recombinant GM-CSF at the dose of 250 mcg/m2 will be given intravenously from day +7 to help white counts recovery. The drug will be diluted in NS at a concentration of at least 10 mcg/ml.
  Drug Information: Sargramostim (Leukine) Formulation: 250 mcg, 500 mcg lyophlized powder for injection

SUMMARY:
The purposes of this study are:

* To examine the engraftment rate in patients receiving in vivo T-cell-depleted G-CSF stimulated bone marrow from partially mismatched related donors.
* To evaluate the incidence and severity of acute and chronic graft-versus-host disease in patients receiving in vivo T-cell-depleted G-CSF stimulated bone marrow from partially mismatched related donors.

DETAILED DESCRIPTION:
This study is a single-arm, non-randomized feasibility study. Patients meeting the criteria for this study will be entered sequentially until completion or closure of the study. Early stopping rules will be employed to ascertain whether an unacceptable rate of toxicity (non-engraftment, and/or acute GVHD) occurs.

Patients will be prepared for transplant through the administration of the following conditioning regimen based on their primary disease:

* Total body irradiation (1400 rads in 8 fractionated doses) and high dose chemotherapy, including cytosine arabinoside, etoposide, and cyclophosphamide. Patients with bone marrow failure syndrome will not receive etoposide in the conditioning regimen.
* Post transplant immunosuppression prophylaxis against acute GVHD will include sequential administration of cyclosporine, methotrexate, basiliximab and mycophenolate.
* The donor will receive 3 daily G-CSF injections prior to marrow harvest starting on day -3. The injections may be initiated by the donor's primary physician prior to donor's arrival, or by the BMT service at Children's Healthcare of Atlanta.
* Patients will receive daily GM-CSF injections (250 mcg/m2) starting from day +7 post transplant until absolute neutrophil count (ANC) is greater than 2,000/µL for three days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hematologic malignancies or bone marrow failure syndrome who are candidates for allogeneic bone marrow transplantation are eligible for this study. Hematologic malignancies indicated for transplantation:

  * Acute lymphoblastic leukemia (ALL) in first remission (with high risk feature), 2nd or greater remission.
  * Acute myeloid leukemia (AML) in first remission (with high risk feature), 2nd or greater remission.
  * Chronic myeloid leukemia (CML) in 2nd chronic phase or accelerated phase.
  * Juvenile myelomonocytic leukemia (JMML).
  * Myelodysplastic syndrome.
  * Biphenotypic leukemia in first (with high risk feature), 2nd or greater remission.
  * Induction failure leukemia.
  * Refractory relapsed leukemia.
  * Bone marrow failure syndrome.
  * Severe aplastic anemia failed immunotherapy.
* Patients who do not have a 6 out of 6 matched related or unrelated donor or 4/6 and 5/6 matched cord blood will be eligible for this study.
* Partially mismatched related donor availability as defined by molecular typing with 3 to 5 HLA matches.
* Patients who are under 22 years of age.

Exclusion Criteria:

* Patients will not be excluded based on sex, racial, or ethnic background.
* Patients will be excluded if they demonstrate significant functional deficits in major organs, which would obviously interfere with successful outcome following bone marrow transplant utilizing the following guidelines.

  * Evidence of active, deep-seated, life-threatening infections for which there is no known effective therapy (certain fungal species, HIV, etc.).
  * Patients who have been treated for infections must have appropriate responses as documented by 2 (two) consecutive negative cultures and/or stable radiographic examinations.
  * Patients who have active central nervous system (CNS) leukemic disease.
* Patients will be excluded if they are women of childbearing potential who are currently pregnant (beta-HCG+) or who are not practicing adequate contraception.
* Patients who have had a previous hematopoietic stem cell transplant will be excluded.
* Donors will be excluded if they are sensitive to E. coli-derived protein.

Max Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2004-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kuang-Yueh Chiang, M.D., Principal Investigator — Children's Healthcare of Atlanta/Emory University
Locations (1):
- Children's Healthcare of Atlanta/Emory University, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Children's Healthcare of Atlanta between January 2005 and December 2013.
Groups:
- Granulocyte Colony Stimulating Factor (G-CSF) Stimulation: Participants with hematologic malignancies or bone marrow failure syndrome received in vivo T-cell depleted granulocyte colony stimulating factor (G-CSF) stimulated bone marrow from a partially mismatched related donor.
Period: Overall Study
Arm/Group | Granulocyte Colony Stimulating Factor (G-CSF) Stimulation
Started | 8
Completed | 4
Not Completed | 4
Not completed — Death | 4

BASELINE CHARACTERISTICS:
Arm/Group | Granulocyte Colony Stimulating Factor (G-CSF) Stimulation
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Engraftment Rate
Description: The number of participants who received in vivo T-cell-depleted G-CSF stimulated bone marrow from partially mismatched related donor who reached engraftment by Day 45.
Time Frame: Day 45
Measure: Number; unit: particpants
Groups:
- Granulocyte Colony Stimulating Factor (G-CSF) Stimulation: Participants received bone marrow from donors who underwent Granulocyte Colony Stimulating Factor (G-CSF) stimulation prior to bone marrow collection.
Arm/Group | Granulocyte Colony Stimulating Factor (G-CSF) Stimulation
Number analyzed (Participants) | 8
particpants | 8

2. Primary Outcome: Incidence of Acute Graft-versus-host Disease
Description: The number of participants diagnosed with new acute graft-versus-host disease (GVHD).
Time Frame: Day 100
Population: Participants who who developed acute GVHD was measured at Day 100 post bone marrow transplant.
Measure: Number; unit: participants
Arm/Group | Granulocyte Colony Stimulating Factor (G-CSF) Stimulation
Number analyzed (Participants) | 8
participants | 6

3. Primary Outcome: Incidence of Chronic Graft-versus-host Disease
Description: The number of participants diagnosed with chronic graft-versus-host disease (GVHD).
Time Frame: Duration of Study (Up to two years)
Population: Participants who survived beyond Day 100 post bone marrow transplant.
Measure: Number; unit: participants
Arm/Group | Granulocyte Colony Stimulating Factor (G-CSF) Stimulation
Number analyzed (Participants) | 6
participants | 2

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the duration of the study and follow up period (up to two years).
Arm/Group | Granulocyte Colony Stimulating Factor (G-CSF) Stimulation
Serious Adverse Events (participants affected / at risk) | 4/8
Other Adverse Events (participants affected / at risk) | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Granulocyte Colony Stimulating Factor (G-CSF) Stimulation (N=8)
Recurrent Disease (Blood and lymphatic system disorders) | 2 (2)
Multi-organ system failure (General disorders) | 2 (2) — Multi-organ system failure was related to severe graft-versus-host disease and resulted in death.

LIMITATIONS AND CAVEATS:
There was a small number of participants and a short follow up time period for this trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes